CLINICAL TRIAL: NCT02381691
Title: Analgesic Effect of Maternal Breast Milk Odor in Preterm Neonates: a Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2012-11; RC12_3630 (Registry Identifier: APHM); 2012-A00360-43 (Other: IDRCB)
Record Dates: First submitted 2015-02-04; First posted 2015-03-06 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Neonates Analgesy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- maternal breast milk odor (Experimental): In the first group "breast milk", venipuncture was performed to the neonate while his mother's milk odor was being diffused.
  Interventions: Other: maternal breast milk odor
- no odor (Placebo Comparator): In a second control group, venipuncture was performed to the neonate with an odorless diffusor.
  Interventions: Other: no odor

INTERVENTIONS:
Other: maternal breast milk odor
  Arms: maternal breast milk odor
Other: no odor
  Arms: no odor

SUMMARY:
Objective : To assess the analgesic effect of maternal breast milk odor in preterm neonates Design : A prospective, randomised, controlled, double blinded, monocentric trial.

Méthods : The neonates were included from 01/01/2012 to 31/12/2014. Inclusion criteria were: neonates fed with their mother breast milk, gestational age between 30 weeks of amenorrhea and 36 weeks + 6 days, a postnatal age ≤ 10 days and a birth weight greater than the 5th percentile according to Olsen curves et al. They also had to be: clinically stable, with 48 hours withdrawal of nasal CPAP, without administration of any analgesic or sedative drug in the last 48 hours and without any underlying disease. The two legal representatives must have signed an informed consent. The study excluded the neonates for whom no video was recorded during the venipuncture.

In the first group "breast milk", venipuncture was performed to the neonate while his mother's milk odor was being diffused. In a second control group, the same gesture was made with an odorless diffusor. The primary outcome was the clinical score assessment PIPP (Premature Infant Pain Profile). The secondary outcomes were the DAN score (Acute Pain of Newborn) and the salivary cortisol level.

ELIGIBILITY:
Inclusion Criteria:

* neonates fed with their mother breast milk,
* gestational age between 30 weeks of amenorrhea and 36 weeks + 6 days,
* postnatal age ≤ 10 days
* birth weight greater than the 5th percentile according to Olsen curves et al.
* clinically stable, with 48 hours withdrawal of nasal CPAP, without administration of any analgesic or sedative drug in the last 48 hours and without any underlying disease
* the two legal representatives must have signed an informed consent.

Exclusion Criteria:

* neonates for whom no video was recorded during the venipuncture

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
clinical score assessment PIPP (Premature Infant Pain Profile) | 20 minutes

SECONDARY OUTCOMES:
DAN score (Acute Pain of Newborn) | 20 minutes
salivary cortisol level | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Desalbres Urielle, Study Director — APHM
Locations (1):
- Assistance Publique des Hopitaux de Marseille, Marseille, France